CLINICAL TRIAL: NCT02237521
Title: The Effect of the Incretin Hormones on the Endocrine Pancreatic Function During Hyperglycemia in End-stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Bo Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, MD DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-2-2014-021
Record Dates: First submitted 2014-08-29; First posted 2014-09-11 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: End-stage Renal Disease
Keywords: Incretin hormones; End-stage renal disease; ESRD; GLP-1; GIP; Insulin; Glucagon
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance | interventions — Arginine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- End-stage renal disease: Patients with normal glucose tolerance and end-stage renal disease
  Interventions: Other: Eu- and hyperglycemic clamp; Other: Arginine test
- Controls: Healthy controls with normal kidney function and normal glucose tolerance
  Interventions: Other: Eu- and hyperglycemic clamp; Other: Arginine test

INTERVENTIONS:
Other: Eu- and hyperglycemic clamp — Eu- and hyperglycemic clamp with concomitant infusion of the natural occurring hormones glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic peptide (GIP) or placebo along with stable glucose isotope infusion to measure the effects of the incretins.
Other: Arginine test — Bolus infusion of the natural occurring amino acid arginine to measure the ability to increase the secretion of insulin and glucagon

SUMMARY:
Patients with end-stage renal disease (ESRD) have a high prevalence of impaired glucose metabolism. The pathophysiological cause is uncertain, but disturbances in the secretion, elimination and effect of glucagon, insulin and the two incretin hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP), probably play important roles. Our research group has previously found that dialysis patients without type 2 diabetes mellitus (T2DM) have a reduced incretin effect and an inability to suppress glucagon after a meal - two early pathophysiological characteristics of patients with T2DM and normal kidney function.

The aim of the project is to provide a detailed description of the mechanisms underlying the (patho)physiological effects of the incretin hormones in patients with ESRD. We plan to investigate the above mentioned disturbances during fasting and hyperglycaemic conditions using incretin infusions during glucose clamping. Furthermore, stable isotopic tracers will be used to determine the effect of the incretin hormones on the endogenous glucose handling.

We hypothesise that the effects of the incretin hormones in ESRD will be reduced in respect to healthy control subjects.

DETAILED DESCRIPTION:
The effect of the incretin hormones on the endocrine pancreatic function in a uremic environment will be explored during fasting and hyperglycemic conditions in three randomised examination days.

At a preceding screening day, an oral glucose tolerance test (OGTT) and a dual energy x-ray absorptiometry (DXA) scan will be performed to determine glucose tolerance and the distribution of muscle and adipose tissue. The study will be carried out on three separate days differing with respect to the hormones infused: GLP-1, GIP or placebo (saline) which are double blinded. The patients will meet from an overnight fast and an infusion of one of the hormones is initiated. At the same time labeled glucose will be infused to determine the endogenous hepatic glucose production. A glucose infusion is adjusted according to frequent plasma glucose measurements to maintain fasting glucose level. After 2 hours a steady state of the tracer is achieved and a 2 hour hyperglycemic clamp, 3 mmol/l above fasting glucose concentration will be started. The tracer infusions are continued during the hyperglycemia. After the 4 hour clamp an arginine bolus will be administered to measure the ability to increase the secretion of insulin and glucagon.

ELIGIBILITY:
Inclusion Criteria (End-stage renal disease):

* Chronic hemodialysis-dependent uremia in more than 3 months

Inclusion Criteria (Healthy controls):

* Normal kidney function

Exclusion Criteria:

* Fasting plasma glucose ≥ 6.1 mmol/l
* 2h plasma glucose ≥ 7.8 after ingestion of 75 grams of glucose
* Admittance to a hospital
* Anemia (Hb < 6.0 mmol/l)
* Ongoing treatment with drugs interfering with glucose metabolism including steroids and calcineurin inhibitors
* Bowel resection or any other large abdominal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. End-stage renal disease patients receiving chronic hemodialysis treatments
  2. Healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
The effect of GLP-1 and GIP on insulin response during hyperglycemia between groups | Average during the last 2 hours of each examination day. Blood samples are collected at time 122, 124, 126, 130, 210, 225 and 240 minutes
  Average plasma insulin concentrations during hyperglycemia

SECONDARY OUTCOMES:
The effect of GLP-1 and GIP on insulin, glucagon and endogenous glucose production during euglycemia | Average during the first 2 hours of each examination day. Blood samples are collected at time 90, 105 and 120 minutes
  Average plasma insulin and glucagon concentrations as well as glucose rate of appearance during euglycemia.
The effect of GLP-1 and GIP on early and late phase of insulin, glucagon and endogenous glucose production during hyperglycemia | Averages during the last 2 hours of each examination day. Blood samples are collected at time 122, 124, 126, 130, 210, 225 and 240 minutes
  Average plasma insulin and glucagon concentrations as well as glucose rate of appearance during the first 10 minutes and last 30 minutes of hyperglycemia.
The effect of GLP-1 and GIP on insulin and glucagon response to arginine | Average following ariginine bolus. Blood samples are collected at time 242, 244, 246 and 250 minutes
  Average plasma insulin and glucagon concentrations 10 minutes following arginine bolus at the end of the examination.
The effect of GLP-1 and GIP on the peripheral glucose handling | Average during the first 4 hours of each examination day. Blood samples are collected at 5-15 minutes interval from time 0 to time 240 minutes
  Average glucose infusion rate during both euglycemia (the first 2 hours) and hyperglycemia (the last 2 hours).
The effect of GLP-1 and GIP on potassium concentrations during euglycemia | Average during the first 2 hours of each examination day. Blood samples are collected at time 30, 60, 90 and 120 minutes
  Average plasma potassium concentrations during euglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Morten B Jørgensen, MD, Principal Investigator — Department of Nephrology, Rigshospitalet
Locations (1):
- Department of Nephrology, Rigshospitalet, Copenhagen, Denmark